CLINICAL TRIAL: NCT06127290
Title: HIV Resistance, Molecular Epidemiology and New Treatment Strategies in the Eastern European Region and in Russia
Status: Recruiting | Type: Observational
Sponsor: Euresist Network GEIE (Other)
Collaborators: Karolinska Institutet (Other); University of Siena (Other); University Hospital of Cologne (Other); Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Other Study IDs: CARE4ART
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-1 patients naive to therapies: HIV-1 patients naive to therapies with sub subtype A6 treated in first line with INSTI

SUMMARY:
Cohort based prospective monitoring of the spread of HIV drug resistance during a phase when new anti-HIV drugs are introduced.

DETAILED DESCRIPTION:
The patient cohort that has been set up includes both viral sequences and clinical/epidemiological data from diverse geographical regions in Russia and Ukraine, where continued prospective follow-up - both short-term and long-term - is warranted to monitor and investigate drug resistance and its impact on INSTI roll-out. Likewise, continued collection of samples and data is fundamental to study the impact of DRM (Drug Resistance Mutations) in Russia and the Eastern European Region for upcoming new drugs, in order to expand the knowledge and to get a representative pattern.

In particular the promoter aims in the timeframe of 1 year at:

* Cohort based prospective monitoring of the spread of HIV drug resistance during a phase when new anti-HIV drugs are introduced. It requires a long-time follow up to identify any changing PDR (Pre-treatment Drug Resistance) patterns.
* Cohort based prospective exploration of the temporal kinetics of subtypes and sub-subtypes in Russia in order to define the coming molecular epidemiology of HIV-1.
* Expand the description of DRM (natural polymorphisms, pre-existing, acquired and off-target mutations) in a larger number of patients mainly from Russia. The samples and the collected data will be used to study the impact of DRM on the phenotypic sensitivity for INSTI and other already diffused drugs (NRTI/NNRTI).
* Support the implementation and evaluation of the PDR surveillance plan which has been defined in accordance with WHO (World Health Organisation) directives.

ELIGIBILITY:
Inclusion Criteria:

* naïve patients starting 2nd generation INSTI treatment
* first line patients under 2nd generation INSTI treatment with either viral RNA sequence before therapy start, or PBMC available with PBMC sample date not more than 3 years from therapy start date (with reasonably sure history of no failure in the interval from therapy start date to PBMC sample date]).

Exclusion Criteria:

* patients not having a signed informed consent for the EIDB data repository, if required by local/national legislation in order to have data in the common data repository.
* patients not having Signed Informed consent for the present study, if required by local authorities iii) Persons aged < 18 at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prospectively enrolled treatment naïve patients who are put on antiretroviral therapy including 2nd generation INSTI. Random selection from the local HIV database will be made among persons who fulfil the inclusion criteria. Consecutive persons from the list attending outpatient clinic will be enrolled by the treating physician/study nurse.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Viral Load at 1 year | 1 year
  Viral Load after one year from the therapy start or at virological failure

SECONDARY OUTCOMES:
number and types of DRM at baseline | 1 week
  drug resistance mutations at baseline
number and types of DRM1 after 1 year | 1 year
  drug resistance mutations after 1 year or at virological failure

CONTACTS AND LOCATIONS:
Overall Officials: FRANCESCA INCARDONA, Study Chair — Euresist Network GEIE
Locations (4):
- University Hospital of Cologne, Cologne, Germany
- University Hospital of Siena, Siena, Italy
- Pomeranian Medical University Szczecin, Szczecin, Poland
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided